CLINICAL TRIAL: NCT01125930
Title: Investigation of the Topical Retinoid, Atralin Gel 0.05% for the Treatment of Erythematotelangiectatic Rosacea
Brief Title: Atralin Gel for the Treatment of Rosacea
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to slow recruitment and sponsor request study ended early
Sponsor: Lisa E. Maier (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lisa E. Maier, Assistant Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Derm 616
Record Dates: First submitted 2010-05-13; First posted 2010-05-19 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Rosacea
Keywords: rosacea; tretinoin; atralin
MeSH Terms: conditions — Rosacea | interventions — Atralin Gel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle gel (Placebo Comparator): Topical gel that does not contain active drug. The gel will be applied initially 3 times per week to the face. If no irritation seen at follow up visit, the investigator will consider increasing the frequency of use. This topical medication will not be applied more than once daily. If there is irritation, the subject will be asked to decrease frequency of use.
  Interventions: Drug: vehicle gel
- Atralin gel (Active Comparator): Topical Atralin gel will be applied initially 3 times per week to the face. If no irritation seen at follow up visit, the investigator will consider increasing the frequency of use. This topical medication will not be applied more than once daily. If there is irritation, the subject will be asked to decrease frequency of use. This drug will be used for the duration of the study.
  Interventions: Drug: Atralin gel

INTERVENTIONS:
Drug: vehicle gel — Topical gel that does not contain active drug. The gel will be applied initially 3 times per week to the face. If no irritation seen at follow up visit, the investigator will consider increasing the frequency of use. This topical medication will not be applied more than once daily. If there is irritation, the subject will be asked to decrease frequency of use.
  Arms: Vehicle gel
Drug: Atralin gel — Topical Atralin gel will be applied initially 3 times per week to the face. If no irritation seen at follow up visit, the investigator will consider increasing the frequency of use. This topical medication will not be applied more than once daily. If there is irritation, the subject will be asked to decrease frequency of use. This drug will be used for the duration of the study.
  Arms: Atralin gel

SUMMARY:
Erythematotelangiectatic rosacea is a type of rosacea that causes a red face often with frequent flushing, topical sensitivity and prominent blood vessels. We think that long term damage to skin from the sun (photodamage) may play a role in causing this type of rosacea. Tretinoin is a topical medication that is known to improve photodamage. We want to find out if Atralin (tretinoin 0.05%) Gel used for up to 46 weeks will improve erythematotelangiectatic rosacea (ETR).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age and older of any race.
2. Clinical diagnosis of mild to moderate erythematotelangiectatic facial rosacea based on physician evaluation.
3. Willing and able to understand and sign informed consent.
4. Able to complete study and comply with study procedures.

Exclusion Criteria:

1. Severe self reported facial sensitivity
2. History of allergy to fish
3. Severe sun sensitivity
4. Severe erythematotelangiectatic rosacea requiring systemic treatment
5. Papulopustular, Ocular-only, Phymatous rosacea, Steroid rosacea, pyoderma faciale
6. Unwilling to undergo facial biopsies
7. Concomitant use of medications that are reported to exacerbate rosacea, such as topical and systemic steroids
8. Use of topical rosacea treatments in the past 2 weeks.
9. Use of systemic antibiotics in the past 4 weeks.
10. Use of systemic retinoids within the past 6 months.
11. Use of topical retinoids within the past 3 months
12. Use of laser or light based rosacea treatments within the past 2 months.
13. Cosmetic procedures (e.g., superficial chemical peels, exfoliation or microdermabrasion of the face) within the past two months
14. Use of topical anti-aging medications including alpha hydroxy acids, salicylic acid, beta-hydroxy acid, vitamin A, vitamin E, ascorbic acid
15. Other dermatologic conditions that require the use of interfering topical or systemic therapy or that might interfere with study assessments.
16. Clinically significant abnormal findings or conditions (other than rosacea), which might, in the opinion of the Investigator, interfere with study evaluations or pose a risk to subject safety during the study.
17. If female, Subjects who are either of non-child bearing potential (defined as postmenopausal -absence of menstrual bleeding for 1 year - or as having undergone bilateral tubal ligation, hysterectomy or bilateral ovariectomy) or, if of childbearing potential, Subjects who have had a negative urine pregnancy test at the beginning of the study, and have agreed to practice appropriate birth-control to prevent pregnancy during the study.(The type and dose of birth control must have been stable for at least 2 months prior to study entry and not be expected to change during the study).
18. Subjects who are lactating.
19. Use of any investigational therapy within the past 4 weeks.
20. Known hypersensitivity or previous allergic reaction to retinoids
21. Carcinoid, Pheochromocytoma or other systemic flushing causes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa E Maier, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Pelle MT, Crawford GH, James WD. Rosacea: II. Therapy. J Am Acad Dermatol. 2004 Oct;51(4):499-512; quiz 513-4. doi: 10.1016/j.jaad.2004.03.033. PMID 15389184
- [Background] Ertl GA, Levine N, Kligman AM. A comparison of the efficacy of topical tretinoin and low-dose oral isotretinoin in rosacea. Arch Dermatol. 1994 Mar;130(3):319-24. PMID 8129410
- [Background] Vienne MP, Ochando N, Borrel MT, Gall Y, Lauze C, Dupuy P. Retinaldehyde alleviates rosacea. Dermatology. 1999;199 Suppl 1:53-6. doi: 10.1159/000051380. PMID 10473962

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle Gel | Atralin Gel
Started | 22 | 46
Completed | 21 | 36
Not Completed | 1 | 10
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Gel | Atralin Gel | Total
Number analyzed (Participants) | 22 | 46 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.00 (11.24) | 56.09 (11.58) | 55.74 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 39 | 54
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian, European descent | 22 | 43 | 65
  Caucasian, non-European descent | 0 | 2 | 2
  Middle Eastern | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 46 | 68

OUTCOME MEASURES:

1. Primary Outcome: Severity of Erythematotelangiectatic Rosacea Signs: Redness (Non Transient Erythema)
Description: Severity of erythematotelangiectatic rosacea signs will be measured by taking into account the following: redness, telangiectasia, facial edema, dry skin
Time Frame: 24 weeks
Population: Last Observation Carried Forward (LOCF), Complete-Case Intent-to-Treat (ITT) Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel | Atralin Gel
Number analyzed (Participants) | 21 | 36
participants
  None | 0 | 0
  Mild Erythema | 12 | 22
  Moderate Erythema | 9 | 13
  Marked Erythema | 0 | 1
  Deep Erythema | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons were done at the Week 24 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess redness; Test type: Superiority or Other; p = 0.93, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

2. Primary Outcome: Severity of Erythematotelangiectatic Rosacea Signs: Telangiectasia
Description: as for outcome 1
Time Frame: 24 weeks
Population: LOCF, Complete-Case ITT population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel | Atralin Gel
Number analyzed (Participants) | 21 | 36
participants
  None | 1 | 0
  Mild | 10 | 22
  Moderate | 10 | 13
  Severe | 0 | 1
Statistical Analysis 1: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons were done at the Week 24 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess telangiectasia; Test type: Superiority or Other; p = 0.79, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

3. Secondary Outcome: Quality of Life
Description: The Dermatology Life Quality Index (DLQI) questionnaire was given at each visit. It involves 10 questions that relate to symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. The total DLQI score is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: 2, 6, 12, 18, 24 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Vehicle Gel at Week 2; Vehicle Gel at Week 6; Vehicle Gel at Week 12; Vehicle Gel at Week 18; Vehicle Gel at Week 24: Vehicle gel: Topical gel that does not contain active drug. The gel will be applied initially 3 times per week to the face. If no irritation seen at follow up visit, the investigator will consider increasing the frequency of use. This topical medication will not be applied more than once daily. If there is irritation, the subject will be asked to decrease frequency of use.
- Atralin Gel at Week 2; Atralin Gel at Week 6; Atralin Gel at Week 12; Atralin Gel at Week 18; Atralin Gel at Week 24: Atralin gel: Topical Atralin gel will be applied initially 3 times per week to the face. If no irritation seen at follow up visit, the investigator will consider increasing the frequency of use. This topical medication will not be applied more than once daily. If there is irritation, the subject will be asked to decrease frequency of use. This drug will be used for the duration of the study.
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18 | Vehicle Gel at Week 24 | Atralin Gel at Week 24
Number analyzed (Participants) | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36
units on a scale | 2.62 (3.01) | 2.28 (2.31) | 2.19 (2.36) | 2.44 (2.21) | 1.95 (2.25) | 2.03 (1.92) | 1.52 (1.63) | 2.14 (2.26) | 1.43 (1.60) | 2.14 (2.43)
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparisons were done at the Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other; Test type: Superiority or Other; p = 0.94, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values to address non-normality of data
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparisons were done at the Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other; Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values to address non-normality of data
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparisons were done at the Week 12 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other; Test type: Superiority or Other; p = 0.66, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values to address non-normality of data
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparisons were done at the Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other; Test type: Superiority or Other; p = 0.38, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values to address non-normality of data
Statistical Analysis 5: Comparison: Vehicle Gel at Week 24 vs Atralin Gel at Week 24; Group comparisons were done at the Week 24 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other; Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values to address non-normality of data

4. Secondary Outcome: Photodamage
Description: Photodamage was measured at baseline and Week 24 visits using the nine point Hamilton-Griffiths Photoaging Score categories. The categories were developed using photographs of subject representing grades of photodamge from none (0) to severe (8). A direct comparison is made between the subject and the photographic standards. If an exact match cannot be made, the interstandard scores (1, 3, 5, 7) are used.
Time Frame: 24 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel | Atralin Gel
Number analyzed (Participants) | 21 | 36
participants
  Score of 0, No Photo Damage | 0 | 0
  Score of 1, Mild Photo Damage, < score of 2 | 3 | 1
  Score of 2, Mild Photo Damage | 5 | 11
  Score of 3, Mild Photo Damage, > score of 2 | 4 | 12
  Score of 4, Moderate Photo Damage | 5 | 9
  Score of 5, Moderate Photo Damage, > score of 4 | 2 | 2
  Score of 6, Moderate/Severe Photo Damage | 2 | 1
  Score of 7, Severe Photo Damage, < score of 8 | 0 | 0
  Score of 8, Severe Photo Damage | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons were done at the Week 24 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess photodamage; Test type: Superiority or Other; p = 0.87, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

5. Secondary Outcome: Signs of Other Rosacea Subtypes: Ocular Manifestations of Rosacea
Description: Signs of other rosacea subtypes using rosacea clinical scores: ocular manifestations of rosacea
Time Frame: 2, 6, 12, 18 and 24 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18 | Vehicle Gel at Week 24 | Atralin Gel at Week 24
Number analyzed (Participants) | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36
participants
  None | 18 | 32 | 19 | 31 | 18 | 32 | 19 | 32 | 19 | 34
  Mild | 3 | 4 | 2 | 4 | 3 | 4 | 2 | 4 | 1 | 2
  Moderate | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparisons were done at the Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess ocular manifestations of rosacea; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparisons were done at the Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess ocular manifestations of rosacea; Test type: Superiority or Other; p = 0.62, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparisons were done at the Week 12 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess ocular manifestations of rosacea; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney); Wilcoxon rank-sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparisons were done at the Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess ocular manifestations of rosacea; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 5: Comparison: Vehicle Gel at Week 24 vs Atralin Gel at Week 24; Group comparisons were done at the Week 24 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess ocular manifestations of rosacea; Test type: Superiority or Other; p = 0.45, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

6. Secondary Outcome: Signs of Other Rosacea Subtypes: Phymatous Changes of Rosacea
Description: Signs of other rosacea subtypes using rosacea clinical scores: phymatous changes of rosacea
Time Frame: 2, 6, 12, 18 and 24 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18 | Vehicle Gel at Week 24 | Atralin Gel at Week 24
Number analyzed (Participants) | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36
participants
  None | 21 | 34 | 21 | 34 | 21 | 34 | 21 | 34 | 21 | 35
  Mild | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 1
  Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparisons were done at the Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess phymatous changes of rosacea; Test type: Superiority or Other; p = 0.53, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparisons were done at the Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess phymatous changes of rosacea; Test type: Superiority or Other; p = 0.53, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparisons were done at the Week 12 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess phymatous changes of rosacea; Test type: Superiority or Other; p = 0.53, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparisons were done at the Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess phymatous changes of rosacea; Test type: Superiority or Other; p = 0.53, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 5: Comparison: Vehicle Gel at Week 24 vs Atralin Gel at Week 24; Group comparisons were done at the Week 24 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess phymatous changes of rosacea; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

7. Secondary Outcome: Signs of Other Rosacea Subtypes: Papulopustular
Description: Signs of other rosacea subtypes includes papulopustular, inflammatory papule count
Time Frame: 2, 6, 12, 18, 24 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Mean (Standard Deviation); unit: inflammatory papule
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18 | Vehicle Gel at Week 24 | Atralin Gel at Week 24
Number analyzed (Participants) | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36
inflammatory papule | 0.19 (0.51) | 0.25 (0.73) | 0.14 (0.48) | 0.28 (0.66) | 0.43 (0.87) | 0.50 (1.59) | 0.48 (0.87) | 0.64 (1.59) | 0.38 (0.67) | 1.03 (2.69)
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values to address non-normality of data
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.41, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values to address non-normality of data
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.66, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values to address non-normality of data
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values to address non-normality of data
Statistical Analysis 5: Comparison: Vehicle Gel at Week 24 vs Atralin Gel at Week 24; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.80, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values to address non-normality of data

8. Secondary Outcome: Molecular Markers of Inflammation
Description: These will be evaluated from skin biopsies from some subjects at baseline and final evaluation at 24 weeks. Gene expression data were normalized and presented as fold change from baseline to week 24 visit. Markers of inflammation include Tachykinin 1 (TAC1), CXC Motif Receptor 4 (CXCR4), CXC Motif Ligand 12 (CXCL12), and Tumor Necrosis Factor Alpha (TNFa).
Time Frame: 24 weeks
Population: ITT Population that completed baseline and Week 24 biopsies
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Vehicle Gel | Atralin Gel
Number analyzed (Participants) | 7 | 9
fold change
  TAC1 Fold Change Score | 2.91 (1.94) | 0.87 (0.90)
  CXCR4 Fold Change Score | 1.39 (1.18) | 1.88 (1.81)
  CXCL12 Fold Change Score | 1.10 (0.80) | 1.20 (0.59)
  TNFa Fold Change Score | 1.24 (0.84) | 1.17 (0.97)
Statistical Analysis 1: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons of TAC1 at Week 24 visit were made using fold change data; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons of CXCR4 at Week 24 visit were made using fold change data; Test type: Superiority or Other; p = 0.35, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons of CXCL12 at Week 24 visit were made using fold change data; Test type: Superiority or Other; p = 0.68, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons of TNFa at Week 24 visit were made using fold change data; Test type: Superiority or Other; p = 0.76, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

9. Secondary Outcome: Molecular Evidence of Photodamage
Description: These will be evaluated from skin biopsies from some subjects at baseline and final evaluation at 24 weeks. Gene expression data were normalized and presented as fold change from baseline to week 24 visit. Markers of photodamage include Collagen 1 (COL-1), Collagen 3 (COL-3), Matrix Metalloproteinase 1 (MMP1), Matrix Metalloproteinase 3 (MMP3), and Matrix Metalloproteinase 9 (MMP9).
Time Frame: 24 weeks
Population: ITT Population that completed baseline and week 24 biopsies
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Vehicle Gel | Atralin Gel
Number analyzed (Participants) | 7 | 9
fold change
  COL-1 Fold Change Score | 1.50 (1.09) | 1.17 (0.65)
  COL-3 Fold Change Score | 1.39 (0.77) | 1.04 (0.63)
  MMP1 Fold Change Score | 1.44 (1.28) | 0.83 (0.60)
  MMP3 Fold Change Score | 2.87 (3.58) | 0.69 (0.64)
  MMP9 Fold Change Score | 2.53 (4.16) | 1.67 (1.60)
Statistical Analysis 1: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons of COL-1 at Week 24 visit were made using fold change data; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons of COL-3 at Week 24 visit were made using fold change data; Test type: Superiority or Other; p = 0.25, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons of MMP-1 at Week 24 visit were made using fold change data; Test type: Superiority or Other; p = 0.41, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons of MMP-3 at Week 24 visit were made using fold change data; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 5: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons of MMP-9 at Week 24 visit were made using fold change data; Test type: Superiority or Other; p = 0.61, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

10. Secondary Outcome: Severity of Erythematotelangiectatic Signs: Non-Transient Erythema (Redness)
Description: Severity of erythematotelangiectatic signs include redness (non-transient erythema), telangiectasia, facial edema, and dry skin.
Time Frame: 2, 6, 12, 18 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18
Number analyzed (Participants) | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36
participants
  None | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0
  Mild Erythema | 11 | 18 | 11 | 16 | 12 | 20 | 11 | 23
  Moderate Erythema | 10 | 17 | 9 | 18 | 8 | 14 | 9 | 11
  Marked Erythema | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2
  Deep Erythema | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparisons were done at the Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess redness; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparisons were done at the Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess redness; Test type: Superiority or Other; p = 0.44, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparisons were done at the Week 12 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess redness; Test type: Superiority or Other; p = 0.41, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparisons were done at the Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess redness; Test type: Superiority or Other; p = 0.94, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

11. Primary Outcome: Severity of Erythematotelangiectatic Rosacea Signs: Facial Edema
Description: as for outcome 1
Time Frame: 24 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel | Atralin Gel
Number analyzed (Participants) | 21 | 36
participants
  None | 21 | 31
  Mild | 0 | 5
  Moderate | 0 | 0
  Severe | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons were done at the Week 24 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess facial edema; Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

12. Primary Outcome: Severity of Erythematotelangiectatic Rosacea Signs: Dry Skin
Description: as for outcome 1
Time Frame: 24 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel | Atralin Gel
Number analyzed (Participants) | 21 | 36
participants
  None | 13 | 16
  Slight Flaking | 7 | 12
  Moderate Flaking/Scaling | 1 | 8
  Marked Scaling/Fissuring | 0 | 0
  Severe Scaling/Fissuring | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons were done at the Week 24 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess dry skin; Test type: Superiority or Other; p = 0.13, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

13. Primary Outcome: Severity of Erythematotelangiectatic Rosacea Symptoms: Self-Reported Presence of Flushing
Description: Flushing is defined as a temporary redness of the face, neck and chest. Subjects were asked to choose the best answer that applied to them in response to the questions "Do you have flushing?".
Time Frame: 24 weeks
Population: LOCF, Complete Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel | Atralin Gel
Number analyzed (Participants) | 21 | 36
participants
  Yes | 19 | 33
  No | 2 | 3
Statistical Analysis 1: Comparison: Vehicle Gel vs Atralin Gel; Group comparison at Week 24 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other; Test type: Superiority or Other; p = 1.00, Fisher Exact

14. Primary Outcome: Severity of Erythematotelangiectatic Rosacea Symptoms: Self-Reported Facial Burning
Description: Severity of erythematotelangiectatic rosacea symptoms was assessed by asking subjects to rate the facial burning feature of their rosacea.
Time Frame: 24 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel | Atralin Gel
Number analyzed (Participants) | 21 | 36
participants
  None | 15 | 28
  Mild | 6 | 7
  Moderate | 0 | 1
  Severe | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons were done at the Week 24 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess self-reported facial burning; Test type: Superiority or Other; p = 0.75, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

15. Primary Outcome: Severity of Erythematotelangiectatic Rosacea Symptoms: Self-Reported Facial Stinging
Description: Severity of erythematotelangiectatic rosacea symptoms was assessed by asking subjects to rate the Facial Stinging feature of their rosacea.
Time Frame: 24 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel | Atralin Gel
Number analyzed (Participants) | 21 | 36
participants
  None | 17 | 27
  Mild | 4 | 8
  Moderate | 0 | 1
  Severe | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons were done at the Week 24 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess self-reported facial stinging; Test type: Superiority or Other; p = 0.68, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

16. Primary Outcome: Severity of Erythematotelangiectatic Rosacea Symptoms: Self-Reported Assessment of Product
Description: Severity of erythematotelangiectatic rosacea symptoms was assessed by asking subjects to give an overall self-assessment of product tolerance.
Time Frame: 24 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel | Atralin Gel
Number analyzed (Participants) | 21 | 36
participants
  Strongly like product | 2 | 8
  Like product | 7 | 7
  Neutral | 9 | 16
  Dislike product | 3 | 5
  Strongly dislike product | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel vs Atralin Gel; Group comparisons were done at the Week 24 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an overall self-assessment of product tolerance; Test type: Superiority or Other; p = 0.77, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

17. Secondary Outcome: Severity of Erythematotelangiectatic Signs: Telangiectasia
Description: as for outcome 10
Time Frame: 2, 6, 12, 18 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18
Number analyzed (Participants) | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36
participants
  None | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
  Mild | 7 | 17 | 9 | 19 | 10 | 20 | 10 | 21
  Moderate | 14 | 18 | 11 | 16 | 10 | 15 | 10 | 14
  Severe | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparisons were done at the Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess telangiectasia; Test type: Superiority or Other; p = 0.41, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparisons were done at the Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess telangiectasia; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparisons were done at the Week 12 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess telangiectasia; Test type: Superiority or Other; p = 0.96, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparisons were done at the Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess telangiectasia; Test type: Superiority or Other; p = 0.91, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

18. Secondary Outcome: Severity of Erythematotelangiectatic Signs: Facial Edema
Description: as for outcome 10
Time Frame: 2, 6, 12, 18 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18
Number analyzed (Participants) | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36
participants
  None | 21 | 33 | 21 | 33 | 21 | 31 | 21 | 32
  Mild | 0 | 2 | 0 | 3 | 0 | 5 | 0 | 4
  Moderate | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparisons were done at the Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess facial edema; Test type: Superiority or Other; p = 0.29, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparisons were done at the Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess facial edema; Test type: Superiority or Other; p = 0.29, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparisons were done at the Week 12 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess facial edema; Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparisons were done at the Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess facial edema; Test type: Superiority or Other; p = 0.29, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

19. Secondary Outcome: Severity of Erythematotelangiectatic Signs: Dryness/Irritation
Description: as for outcome 10
Time Frame: 2, 6, 12, 18 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18
Number analyzed (Participants) | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36
participants
  None | 8 | 13 | 13 | 13 | 12 | 10 | 13 | 14
  Slight Flaking | 12 | 17 | 7 | 19 | 8 | 18 | 6 | 14
  Moderate Flaking/Scaling | 1 | 5 | 1 | 3 | 1 | 7 | 2 | 8
  Marked Scaling/Fissuring | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Severe Scaling/Fissuring | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparisons were done at the Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess dry skin; Test type: Superiority or Other; p = 0.54, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparisons were done at the Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess dry skin; Test type: Superiority or Other; p = 0.06, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparisons were done at the Week 12 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess dry skin; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparisons were done at the Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess dry skin; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

20. Secondary Outcome: Severity of Erythematotelangiectatic Rosacea Symptoms: Self-Reported Presence of Flushing
Description: Evaluation of erythematotelangiectatic rosacea symptoms includes subject reporting of flushing, burning, stinging, topical product intolerance
Time Frame: 2, 6, 12, 18 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18
Number analyzed (Participants) | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36
participants
  Yes | 17 | 34 | 18 | 32 | 18 | 32 | 18 | 34
  No | 4 | 2 | 3 | 4 | 3 | 4 | 3 | 2
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparison at Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have different values than the other; Test type: Superiority or Other; p = 0.18, Fisher Exact
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparison at Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have different values than the other; Test type: Superiority or Other; p = 0.70, Fisher Exact
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparison at Week 12 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have different values than the other; Test type: Superiority or Other; p = 0.70, Fisher Exact
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparison at Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have different values than the other; Test type: Superiority or Other; p = 0.35, Fisher Exact

21. Secondary Outcome: Severity of Erythematotelangiectatic Rosacea Symptoms: Self-Reported Facial Burning
Description: as for outcome 20
Time Frame: 2, 6, 12, 18 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18
Number analyzed (Participants) | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36
participants
  None | 16 | 26 | 17 | 24 | 16 | 23 | 16 | 24
  Mild | 3 | 7 | 3 | 10 | 5 | 8 | 5 | 10
  Moderate | 2 | 2 | 1 | 1 | 0 | 5 | 0 | 2
  Severe | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparisons were done at the Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess self-reported facial burning; Test type: Superiority or Other; p = 0.80, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparisons were done at the Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess self-reported facial burning; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparisons were done at the Week 12 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess self-reported facial burning; Test type: Superiority or Other; p = 0.25, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparisons were done at the Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess self-reported facial burning; Test type: Superiority or Other; p = 0.46, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

22. Secondary Outcome: Severity of Erythematotelangiectatic Rosacea Symptoms: Self-Reported Facial Stinging
Description: as for outcome 20
Time Frame: 2, 6, 12, 18 weeks
Population: LOCF, Complete-Case ITT Population
Measure: Number; unit: participants
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18
Number analyzed (Participants) | 21 | 36 | 21 | 36 | 21 | 36 | 21 | 36
participants
  None | 17 | 25 | 19 | 24 | 19 | 26 | 19 | 26
  Mild | 4 | 10 | 2 | 10 | 2 | 9 | 2 | 8
  Moderate | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Severe | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparisons were done at the Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess self-reported facial stinging; Test type: Superiority or Other; p = 0.41, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparisons were done at the Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess self-reported facial stinging; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparisons were done at the Week 12 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess self-reported facial stinging; Test type: Superiority or Other; p = 0.16, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparisons were done at the Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to assess self-reported facial stinging; Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

23. Secondary Outcome: Severity of Erythematotelangiectatic Rosacea Symptoms: Self-Reported Product Assessment
Description: as for outcome 20
Time Frame: 2, 6, 12, 18 weeks
Population: LOCF, Complete-Case ITT Population One subject did not complete the product assessment questionnaire at week 2 visit.
Measure: Number; unit: participants
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18
Number analyzed (Participants) | 20 | 36 | 21 | 36 | 21 | 36 | 21 | 36
participants
  Strongly like product | 0 | 3 | 2 | 3 | 2 | 5 | 1 | 7
  Like product | 3 | 8 | 4 | 9 | 4 | 11 | 5 | 9
  Neutral | 17 | 23 | 13 | 20 | 12 | 18 | 13 | 18
  Dislike product | 0 | 2 | 2 | 4 | 2 | 2 | 2 | 2
  Strongly dislike product | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparisons were done at the Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an overall self-assessment of product tolerance; Test type: Superiority or Other; p = 0.36, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparisons were done at the Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an overall self-assessment of product tolerance; Test type: Superiority or Other; p = 0.88, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparisons were done at the Week 12 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an overall self-assessment of product tolerance; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparisons were done at the Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an overall self-assessment of product tolerance; Test type: Superiority or Other; p = 0.17, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

24. Secondary Outcome: Skin Irritation Assessed by Facial Stinging Upon Product Application
Time Frame: 2, 6, 12, 18 weeks
Population: LOCF, Complete-Case ITT Population One subject did not complete the product assessment questionnaire at week 2 visit.
Measure: Number; unit: participants
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18
Number analyzed (Participants) | 20 | 36 | 21 | 36 | 21 | 36 | 21 | 36
participants
  No stinging | 17 | 24 | 20 | 20 | 20 | 25 | 19 | 25
  A little stinging | 3 | 12 | 1 | 15 | 1 | 9 | 2 | 11
  A lot of stinging | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparisons were done at the Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an assessment of skin irritation by facial stinging upon product application; Test type: Superiority or Other; p = 0.21, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparisons were done at the Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an assessment of skin irritation by facial stinging upon product application; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparisons were done at the Week 12 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an assessment of skin irritation by facial stinging upon product application; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparisons were done at the Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an assessment of skin irritation by facial stinging upon product application; Test type: Superiority or Other; p = 0.10, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

25. Secondary Outcome: Skin Irritation Assessed by Facial Itching Upon Product Application
Time Frame: 2, 6, 12, 18 weeks
Population: LOCF, Complete-Case ITT Population One subject did not complete the product assessment questionnaire at week 2 visit.
Measure: Number; unit: participants
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18
Number analyzed (Participants) | 20 | 36 | 21 | 36 | 21 | 36 | 21 | 36
participants
  No itching | 18 | 31 | 21 | 27 | 21 | 30 | 21 | 31
  A little itching | 2 | 5 | 0 | 7 | 0 | 5 | 0 | 4
  A lot of itching | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparisons were done at the Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an assessment of skin irritation by facial itching upon product application; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparisons were done at the Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an assessment of skin irritation by facial itching upon product application; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparisons were done at the Week 12 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an assessment of skin irritation by facial itching upon product application; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparisons were done at the Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an assessment of skin irritation by facial itching upon product application; Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

26. Secondary Outcome: Skin Irritation Assessed by Facial Burning Upon Product Application
Time Frame: 2, 6, 12, 18 weeks
Population: LOCF, Complete-Case ITT Population One subject did not complete the product assessment questionnaire at week 2 visit.
Measure: Number; unit: participants
Arm/Group | Vehicle Gel at Week 2 | Atralin Gel at Week 2 | Vehicle Gel at Week 6 | Atralin Gel at Week 6 | Vehicle Gel at Week 12 | Atralin Gel at Week 12 | Vehicle Gel at Week 18 | Atralin Gel at Week 18
Number analyzed (Participants) | 20 | 36 | 21 | 36 | 21 | 36 | 21 | 36
participants
  No burning | 17 | 28 | 19 | 26 | 20 | 24 | 19 | 29
  A little burning | 3 | 7 | 2 | 10 | 1 | 10 | 2 | 6
  A lot of burning | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Statistical Analysis 1: Comparison: Vehicle Gel at Week 2 vs Atralin Gel at Week 2; Group comparisons were done at the Week 2 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an assessment of skin irritation by facial burning upon product application; Test type: Superiority or Other; p = 0.67, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 2: Comparison: Vehicle Gel at Week 6 vs Atralin Gel at Week 6; Group comparisons were done at the Week 6 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an assessment of skin irritation by facial burning upon product application; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 3: Comparison: Vehicle Gel at Week 12 vs Atralin Gel at Week 12; Group comparisons were done at the Week 21 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an assessment of skin irritation by facial burning upon product application; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values
Statistical Analysis 4: Comparison: Vehicle Gel at Week 18 vs Atralin Gel at Week 18; Group comparisons were done at the Week 18 visit. The null hypothesis that the two groups are the same, was tested against the alternative hypothesis that one group tended to have larger values than the other over the ordinally scaled categories used to provide an assessment of skin irritation by facial burning upon product application; Test type: Superiority or Other; p = 0.42, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test with exact p-values

ADVERSE EVENTS:
Time Frame: Safety assessment was conducted for all subjects at each visit after enrollment in the study. The study duration could range from 24 to 46 weeks.
Arm/Group | Vehicle Gel | Atralin Gel
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/46
Other Adverse Events (participants affected / at risk) | 13/22 | 25/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Gel (N=22) | Atralin Gel (N=46)
Right Hip Osteoarthritis (Surgical and medical procedures) | 0 (0) | 1 (1) — Hip Replacement Surgery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Gel (N=22) | Atralin Gel (N=46)
Tearing of the eyes (Eye disorders) | 0 (0) | 1 (1)
Blurry Vision (Eye disorders) | 1 (1) | 0 (0)
Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Acid GI Reflux (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (8) | 9 (11) — Nasal/Sinus Congestion, Cold, Upper Respiratory Infection
Stomach Flu (Infections and infestations) | 2 (2) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Head Lice (Infections and infestations) | 0 (0) | 1 (1) — Exposure to head lice
Stye (Infections and infestations) | 1 (1) | 0 (0) — Stye of upper eyelid
GI Distress (Infections and infestations) | 1 (1) | 0 (0)
Infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Possible infection of bx
Back Disc Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Back problem (disc) L leg pain
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — R shoulder tendonitis
Arthritis Flare (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Arthritis flare L thumb
Heel Spur (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — L Heel Spur
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Decreased Memory (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety/Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) — Increased hypertension
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) — Nasal/Sinus Drainage, Congestion, Allergies
Asthma Flare (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Irritiated Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) — Facial Irritation, Sunburn
Eczema/Atopic Dermatitis (Skin and subcutaneous tissue disorders) | 2 (3) | 5 (6)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4) — Flare, Development
Papular Inflammatory Flare (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (9)
Nail Disease (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) — Paronychia, Brittle Nails
Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Inflamed Lesion/Cysts (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6) — Inflamed Cyst, Lesion, Bites, Cold Sores
Numbness on Tongue (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination of study due to slow recruitment and sponsor request resulted in smaller number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less